CLINICAL TRIAL: NCT06048172
Title: How Effective and Safe is Trauma Therapy Using Prolonged Exposure for Patients With PTSD and a Comorbid Psychotic Disorder? Treatment Trauma and Psychosis -TEP
Brief Title: Effectiveness of Trauma Therapy Using Prolonged Exposure for Patients With PTSD and a Comorbid Psychotic Disorder
Acronym: TEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medicalschool Hamburg (Other)
Collaborators: Psychiatrische Klinik Lüneburg (Unknown); Regioklinikum Elmshorn (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSH
Record Dates: First submitted 2023-05-15; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Post Traumatic Stress Disorder; PTSD; Psychosis
Keywords: PTSD; schizophrenia; Prolonged Exposure
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Intervention Model Description: Randomised controlled trail (RCT).
Who Masked: Participant
Masking Description: Treatment as usual group compared to intervention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waiting control group (No Intervention): The patients in the treatment-as-usual control group remain on the waiting list for 14 weeks after the baseline measurement. After 14 weeks, they participate in the study diagnostics post-treatment at time point.
- Intervention group (Experimental): In the intervention condition, patients are treated directly after the baseline measurement by Prolonged Exposure in 16 hours of individual therapy. The 16 individual therapy sessions will take place in 1 to 2 sessions per week over a period of 7 to 16 weeks. The individual therapy sessions are videotaped with camera focus on the therapist. Parts of the Prolonged Exposure process (the re-experiencing of the traumatic memory) are recorded on tape, so that the patient can listen to the recording as homework at home. Afterwards, the patients take part in a study diagnostic session.
  Interventions: Behavioral: Prolonged Exposure

INTERVENTIONS:
Behavioral: Prolonged Exposure — In the intervention condition, patients are treated directly after the baseline measurement by Prolonged Exposure in 16 hours of individual therapy. The 16 individual therapy sessions will take place in 1 to 2 sessions per week over a period of 7 to 16 weeks. The individual therapy sessions are videotaped with camera focus on the therapist. Parts of the Prolonged Exposure process (the re-experiencing of the traumatic memory) are recorded on tape, so that the patient can listen to the recording as homework at home. Afterwards, the patients take part in a study diagnostic session.
  Other Names: trauma therapy; PE
  Arms: Intervention group

SUMMARY:
Psychosis patients with comorbid PTSD will be treated with trauma therapy.

DETAILED DESCRIPTION:
This is a monocentric, controlled, prospective, randomised trial. (RCT). The study population is outpatients with psychotic illness and comorbid post-traumatic stress disorder who have applied for outpatient psychotherapy at the psychotherapeutic outpatient clinic (HSA) of the Medical School Hamburg. It will be investigated whether trauma therapy (Prolonged Exposure) reduces PTSD and psychosis symptoms in comparison to the waiting group. The study will be conducted from 01.09.2023 to 30.04.2028. Patients with suitable symptoms should be seen in the psychotherapeutic outpatient (psychotherapeutic consultation hours) at the HSA should be made aware of the study.

In the next step, a detailed diagnosis is made and, if consent is given and the inclusion criteria listed below are met, the patients are enrolled in the study.

The sample size for the longitudinal intent-to-treat (ITT) analysis with a linear mixed model (LMM) was chosen. Models (LMM) was calculated based on a previous RCT (Van den Berg et al., 2016, effect size for PE in CAPS versus waitlist (TAU) d = 0.78, p < 0.001; effect size for PE in paranoia versus waitlist (TAU) d = 0.62, p = .005). ITT analyses with LLM are relatively robust to missing data, despite which we calculate a 20% dropout rate. With an alpha of 0.05; a mean effect size of 0.5, 3 measurement replicates (baseline measurement T0, post-treatment T1, 6-month follow-up after post, T2), we require 28 patients per treatment arm. A total of 56 patients will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a psychotic disorder (F20) or affective disorder with psychotic symptoms(F30) according to DSM-5.
* comorbid post-traumatic stress disorder (PTSD) according to DSM-5 (CAPS-5 score ≥ 23)
* At least 18 years old
* Good knowledge of the German language
* Willingness to participate in randomisation and trauma-focused therapy

Exclusion Criteria:

* Changes in neuroleptic or antidepressant therapy within the last 4 weeks (exclusion of drug effects).
* Any substance dependence with continued use other than nicotine and/or caffeine dependence.
* IQ of 70 or less
* Acute suicidality
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2028-05-17 (Estimated); Study Completion 2028-05-17 (Estimated)

PRIMARY OUTCOMES:
severity of PTSD symptoms | baseline (pre-intervention), post-intervention (after 16 psychotherapy sessions or for waiting group after 4 months) and follow-up (after 6 months)
  Clinical-Administered PTSD Scale for DSM-5 (CAPS, Blake etal., 1998), presence of PTSD and score for severity of PTSD symptoms
Remission of PTSD diagnosis | baseline (pre-intervention), post-intervention (after 16 psychotherapy sessions or for waiting group after 4 months) and follow-up (after 6 months)
  Clinical-Administered PTSD Scale for DSM-5 (CAPS, Blake etal., 1998), presence of PTSD diagnosis (cut-off score lower than 23)

SECONDARY OUTCOMES:
subjective PTSD symptoms | baseline (pre-intervention), post-intervention (after 16 psychotherapy sessions or for waiting group after 4 months) and follow-up (after 6 months)
  sum score of the Posttraumatic Stress Symptom Scale Self-Report (PSSI, Foa et al., 1993), PTSD Di-agnostic Scale (PDS-5, Foa et al., 2013).
severity of psychosis | baseline (pre-intervention), post-intervention (after 16 psychotherapy sessions or for waiting group after 4 months) and follow-up (after 6 months)
  Psychotic Symptom Rating Scales (PSYRATS, Haddock et al.,1991), score for severity of delusions (PSYRATS-DRS) and for severity of auditory hallucinations (PSYRATS-AHRS).
Wellbeing | baseline (pre-intervention), post-intervention (after 16 psychotherapy sessions or for waiting group after 4 months) and follow-up (after 6 months)
  Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS, NHSHealth Scotland, University of Warwick and University of Edinburgh, 2007)

CONTACTS AND LOCATIONS:
Locations (1):
- Medicalschool Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No